CLINICAL TRIAL: NCT06468982
Title: Evidence of the Advantages of Preoperative Intra-aortic Balloon Pump in Surgical Revascularization of Acute Myocardial Infarction
Brief Title: Use of Intra-aortic Balloon Pump Before Surgery for Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ümit arslan, associate professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AÜ-CVS-UA-01
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease; Coronary Bypass Graft Stenosis of Autologous Vessel; Troponin; IABP - Disorder of Intra-Aortic Balloon Pump
Keywords: Acute myocardial infarction; coronary artery bypass surgery; intra-aortic balloon pump; high-sensitivity cardiac troponin I
MeSH Terms: conditions — Coronary Artery Disease | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Intervention Model Description: two groups for patients with acute myocardial infarction scheduled for coronary artery bypass Grafting: Group A with IABP support, and Group B (the control group) without IABP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (IABP support) (Active Comparator): Patients who are receiving intra-aortic balloon pump support during the preoperative period
  Interventions: Device: Intra-aortic Balloon Pump
- Group B (control group; without IABP support) (No Intervention): Patients who did not receive intra-aortic balloon pump support in the preoperative period; control group

INTERVENTIONS:
Device: Intra-aortic Balloon Pump — It will be applied to patients with acute myocardial infarction who have elevated troponin levels and recurrent or persistent chest pain at rest, hemodynamic instability, multivascular disease, left main coronary artery disease, and patients with narrow and/or tortuous coronary artery anatomy in whom PCI has failed or is not applicable.
  Other Names: Datascope Corp. model:The CS300 with IntelliSense combines fiber-optic
  Arms: Group A (IABP support)

SUMMARY:
The optimal timing of surgery in patients with acute myocardial infarction (AMI) and the utilization of preoperative intra-aortic balloon pumps (IABP) in these patients are subjects of ongoing discussion and disagreement. This study aimed to investigate the effects of preoperative IABP on troponin levels, surgical timing, and intraoperative and postoperative outcomes for patients with AMI who undergo coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) is the first treatment for myocardial ischemia; however, if left main coronary artery disease, multivessel disease, or complex architecture disable PCI, 10% of patients may need coronary artery bypass grafting (CABG). Abstinence from surgical reperfusion in patients with acute myocardial infarction (AMI) may be justified due to surgery's 50% mortality rate. An intra-aortic balloon pump (IABP) can help patients who have ongoing ischemia and high cardiac enzymes because it changes the way the heart uses oxygen by increasing coronary blood flow and lowering afterload. Some guidelines do not recommend the use of IABP in patients with AMI except for mechanical complications or shock. Nevertheless, it is commonly acknowledged that the specific criteria for employing IABP differ among clinics and are determined by clinical expertise. Patients with AMI who have impaired coronary perfusion and require surgical revascularization can benefit from preoperative intra-aortic balloon pump (IABP) support. This intervention leads to reorganization of coronary perfusion, resulting in a decrease in elevated troponin levels and quicker myocardial recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had acute myocardial infarction and have been decided on coronary surgical revascularization

Exclusion Criteria:

* mechanical complications of Acute Myocardial Infarction (such as a ruptured chordal or ventricular septum)
* peripheral arterial disease
* renal failure
* history of cerebrovascular accident
* acute cardiogenic shock and cardiac arrest
* reoperation and combined operations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ümit Arslan, assoc prof, Principal Investigator — Ataturk University
Locations (2):
- Turkey (Türkiye) (2):
  - Atatürk University, Yakutiye, Erzurum
  - Atatürk University, Erzurum

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were selected based on their participation in a single center's cardiovascular surgery and cardiology council from May 2021 to December 2023. The first participant was enrolled on May 1, 2021 and the last participant was enrolled on December 31,2023.
Groups:
- Group A (IABP Support): Patients who are receiving intra-aortic balloon pump support during the preoperative period
  Intra-aortic Balloon Pump: in patients with acute myocardial infarction involving elevated troponin levels and recurrent or persistent chest pain at rest, hemodynamic instability, multivessel disease, left main coronary artery disease, and narrow and/or tortuous coronary artery anatomy in which PCI has failed or is not feasible.
Period: Overall Study
Arm/Group | Group A (IABP Support) | Group B (Control Group; Without IABP Support)
Started | 64 | 92
Completed | 64 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (IABP Support) | Group B (Control Group; Without IABP Support) | Total
Number analyzed (Participants) | 64 | 92 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] — Group A had an age range of 39 to 82 years, while Group B had an age range of 35 to 84 years.
  years | 63.1 (8.9) | 65.2 (8.1) | 64.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants] — The study included patients who underwent coronary artery bypass graft surgery, regardless of gender.
  Participants
    Female | 17 | 67 | 84
    Male | 47 | 25 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 64 | 92 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
High sensitive cardiac troponin-I levels [Mean (Standard Deviation); unit: ng/mL] — High-sensitivity cardiac troponin(hs-cTI) is used to diagnose for heart attacks. hs-cTI levels were quantified using a standardized electrochemiluminescence immunoassay. The limit of detection and the 99th percentile upper reference limit were determined based on the guidelines. Reference values were accepted as 0-0.04 ng/mL for both genders. The hs-cTI levels reported correspond to the values measured on the day of patient admission to our clinic. In Group A, the levels ranged from 5.4 to 83.6 ng/mL and in Group B,ranged from 1.1 to 92.5 ng/mL.
  ng/mL | 29.2 (20.5) | 17.3 (16.6) | 20.4 (18.3)
EuroScore II [Mean (Standard Deviation); unit: Percentage of risk (%)] — EuroSCORE II is a validated risk model with 18 parameters estimating mortality in cardiac surgery (www.euroscore.org). It represents the percentage likelihood of mortality, predicting how many similar patients may die. The scale ranges from 0% to %100. Higher values indicate worse prognosis and higher mortality risk. In this study, EuroSCORE II ranged from 0.5% to 7.4% in Group A and 0.6% to 6.8% in Group B
  Percentage of risk (%) | 2.2 (1.4) | 2 (1.2) | 2.1 (1.2)
Chest pain score [Mean (Standard Deviation); unit: scores on a scale] — he Wong-Baker FACES Pain Rating Scale assesses pain intensity using facial features on a 0-10 scale (0 = No hurt, 10 = Hurts worst). Individuals select the image that best represents their pain level (www.wongbakerfaces.org). In this study, pain scores ranged from 4 to 10 in Group A and from 0 to 8 in Group B.
  scores on a scale | 7.6 (1.8) | 2.3 (1.4) | 5.1 (3.2)
C-reactive protein levels [Mean (Standard Deviation); unit: mg/L (0-5)] — C-reactive protein (CRP) is an acute-phase reactant produced by the liver in response to inflammation. CRP levels elevate during myocardial infarction (MI) primarily due to the inflammatory response triggered by myocardial injury. The normal range for CRP levels is generally considered to be less than 5 mg/L. The CRP levels in participants ranged from 3.2 to 115 mg/L for Group A and from 1.8 to 96 mg/L for Group B.
  mg/L (0-5) | 23.4 (19.8) | 21.7 (16.4) | 22.2 (17.3)
Percentage of glycated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] — HbA1c, also known as glycated hemoglobin, is an important biomarker for assessing glucose control, with elevated levels associated with an increased risk of diabetes-related complications; these levels are expressed as a percentage.(normal range 4.0% to 5.6%) It was measured at 4.0-13.4% in Group A patients and 4.3-12.5% in Group B patients.
  percentage of glycated hemoglobin | 7.4 (2.3) | 6.7 (1.9) | 6.8 (2.1)
Left ventricular ejection fraction [Mean (Standard Deviation); unit: percentage of ejected blood (50-65%)] — Ejection fraction (EF) is a measurement that indicates the percentage of blood that is pumped out of the heart's left ventricle during each contraction, relative to the total volume of blood in the ventricle. It serves as a critical indicator of cardiac function, and is commonly used in the assessment of heart conditions, such as heart failure, with normal values typically ranging from 55% to 65%. The ejection fraction (EF) range in both groups of participants was 30% to 60%.
  percentage of ejected blood (50-65%) | 44.9 (7.7) | 47.9 (7.0) | 47.1 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: High-Sensitivity Cardiac Troponin Levels From Days 0-7
Description: Daily repeated measurements of high-sensitivity cardiac troponin (hs-cTnI) on the ng/mL scale were compared between the two groups. The study hypothesizes that hs-cTnI levels decrease more rapidly in participants receiving IABP support compared to those without IABP. This decrease is posited to reflect a myocardial healing process.
Time Frame: 0-7 days
Population: Daily troponin results were recorded for both groups
Measure: Mean (Standard Deviation); unit: ng/mL (0-0.04)
Arm/Group | Group A (IABP Support) | Group B (Control Group; Without IABP Support)
Number analyzed (Participants) | 64 | 92
ng/mL (0-0.04)
  0.days | 29.2 (20.5) | 17.3 (16.6)
  1.days | 23.2 (17.7) | 16.7 (16.3)
  2.days | 15.8 (13.2) | 14.9 (14.8)
  3.days | 9.9 (9.3) | 12.3 (12.6)
  4.days: number analyzed (Participants) | 56 | 92
  4.days | 5.9 (6.2) | 9.5 (12.8)
  5.days: number analyzed (Participants) | 36 | 88
  5.days | 4.4 (4.5) | 6.9 (10)
  6.days: number analyzed (Participants) | 23 | 73
  6.days | 2.3 (2.2) | 5.3 (7.5)
  7.days: number analyzed (Participants) | 9 | 50
  7.days | 1.5 (1.7) | 4.2 (5.6)
Statistical Analysis 1: Comparison: Group A (IABP Support) vs Group B (Control Group; Without IABP Support); After testing for normality, the baseline characteristics of the two groups will be analyzed using the Student's t-test or the Mann-Whitney U-test for continuous variables and the chi-square test or Fisher's exact test for categorical variables. Differences between the intra-aortic balloon pump group and the control group in terms of repeated measurements will be analyzed using mixed ANOVA; Test type: Superiority — To evaluate whether intra-aortic balloon pump catheter support contributes to a more rapid decrease in troponin levels and faster myocardial recovery, daily troponin levels were analyzed using mixed ANOVA; p = 0.05, ANOVA — The p-value was adjusted for multiple comparisons, and the threshold value was set at 0.05; The hypothesis that IABP causes a rapid increase in troponin levels was analyzed using ANOVA, and the p-value was reported

2. Secondary Outcome: In-hospital Mortality
Description: Deaths occurring in the first 30 days after the operation have been defined as mortality.
Time Frame: 0-30 days
Population: The analysis includes patients with acute myocardial infarction undergoing coronary artery bypass grafting (CABG) and follows mortality 0-30 days postoperatively, defined as in-hospital death.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (IABP Support) | Group B (Control Group; Without IABP Support)
Number analyzed (Participants) | 64 | 92
Participants | 4 | 7
Statistical Analysis 1: Comparison: Group A (IABP Support) vs Group B (Control Group; Without IABP Support); The prognostic value of risk factors for in-hospital mortality was evaluated by multivariate logistic regression analysis; Test type: Other; p < 0.05, Wilcoxon (Mann-Whitney); Hazard Ratio, log = 0.55, 95% CI 2-sided [0.38 to 0.78]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the period from the 1st to the 30th postoperative day for each patient who underwent coronary artery bypass grafting surgery
Description: Adverse effects, including neurological complications, atrial fibrillation, low output syndrome, and revision due to bleeding, were recorded among participants in both groups.
Arm/Group | Group A (IABP Support) | Group B (Control Group; Without IABP Support)
All-Cause Mortality (participants affected / at risk) | 4/64 | 7/92
Serious Adverse Events (participants affected / at risk) | 12/64 | 13/92
Other Adverse Events (participants affected / at risk) | 12/64 | 16/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (IABP Support) (N=64) | Group B (Control Group; Without IABP Support) (N=92)
low cardiac output syndrome (Cardiac disorders) | 2 | 5
Neurological complications (Nervous system disorders) | 1 | 4 — cerebrovascular accident; stroke
Surgical revision for bleeding (Blood and lymphatic system disorders) | 9 | 4 — Re-operation due to drainage due to postoperative mediastinal bleeding
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (IABP Support) (N=64) | Group B (Control Group; Without IABP Support) (N=92)
Atrial fibrillation (Cardiac disorders) | 12 | 16

LIMITATIONS AND CAVEATS:
Not using more than one troponin test kit. The Swan-Ganz catheter or cardiac index device cannot be used in every patient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT06468982/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT06468982/ICF_001.pdf